CLINICAL TRIAL: NCT00047099
Title: A Randomized Phase III Trial Comparing FEC-Chemotherapy vs. EC-Doc-Chemotherapy in Patients With Primary Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: LMU-ADEBAR; LMU-ADEBAR; EU-20221
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2002-12

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Goserelin; Tamoxifen; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: goserelin acetate
Drug: tamoxifen citrate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them after surgery may kill any remaining tumor cells following surgery. It is not yet known which combination chemotherapy regimen is more effective in treating breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different combination chemotherapy regimens in treating women who have primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to progression of women with primary breast cancer treated with fluorouracil, epirubicin, and cyclophosphamide vs docetaxel, epirubicin, and cyclophosphamide.
* Compare the overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to metastatic axillary lymph node involvement (4-9 vs 10 or more), hormone receptor status (estrogen and/or progesterone) of the primary tumor (negative vs positive), and timing of adjuvant radiotherapy (intermittently after completion of 50% of chemotherapy vs after completion of all chemotherapy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fluorouracil IV over 10-15 minutes and epirubicin IV over 15 minutes on days 1 and 8 and oral cyclophosphamide on days 1-14. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive epirubicin IV over 15 minutes and cyclophosphamide IV over 1 hour on days 1, 21, 42, and 63 and docetaxel IV over 1 hour on days 84, 105, 126, and 147 in the absence of disease progression or unacceptable toxicity.

Within 21 days after the completion of chemotherapy, patients undergo adjuvant radiotherapy 5 days a week for 5.5 weeks. Alternatively, patients may undergo radiotherapy intermittently after completion of 50% of chemotherapy.

Upon completion of chemotherapy, patients with positive hormone receptor status (estrogen and/or progesterone) receive oral tamoxifen daily for 5 years. Additionally, patients with positive hormone receptor status who are under age 40 receive goserelin subcutaneously every 4 weeks for 2 years.

Quality of life is assessed at baseline, prior to each course of chemotherapy, 4 weeks after completion of chemotherapy, 6 weeks after completion of radiotherapy, and then at 6 months after completion of chemotherapy.

Patients are followed every 3 months for 3 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 446 patients (223 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary epithelial invasive carcinoma of the breast

  * T1-4, N1-2, M0
  * Must have 4 metastatic axillary lymph nodes
* Complete resection of the primary tumor within the past 5 weeks

  * Free of invasive carcinoma with at least 10 lymph nodes removed
* No inflammatory breast cancer
* No distant metastases by chest x-ray, liver ultrasound, and whole body bone scan
* Hormone receptor status:

  * Estrogen and/or progesterone receptor status known

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 32 weeks

Hematopoietic

* WBC at least 3,000/mm3
* Platelet count at least 100,000

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN
* Albumin no greater than 1.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No cardiomyopathy with impaired ventricular function
* No New York Heart Association class III or IV heart disease
* No cardiac arrhythmias influencing LVEF and requiring medication
* No myocardial infarction within the past 6 months
* No angina pectoris within the past 6 months
* No uncontrolled arterial hypertension

Other

* No other primary malignancy except carcinoma in situ of the cervix or adequately treated basal cell skin cancer
* No known hypersensitivity to docetaxel, epirubicin, fluorouracil, cyclophosphamide, or other study medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic or other antineoplastic therapy
* No other concurrent cytotoxic or other antineoplastic therapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 3 weeks since prior investigational agents

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2001-08; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Comparison of time to progression

SECONDARY OUTCOMES:
Overall survival time
Toxicity
Changes in quality of life over time as measured by the EORTC QLQ-C30 and BR23 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sommer, MD, Study Chair — Ludwig-Maximilians - University of Munich
Locations (2):
- Germany (2):
  - I. Frauenklinik und Hebammenschule der Ludwig-Maximillians Universitaet Muenchen, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich

REFERENCES:
- [Result] Janni JW, Sommer H, Rack B, et al.: The ADEBAR trial: final toxicity analysis of a phase III study evaluating the role of docetaxel in the adjuvant therapy of breast cancer patients with extensive lymph node involvement. [Abstract] J Clin Oncol 25 (Suppl 18): A-585, 24s, 2007.
- [Result] Gauger K, Bismarck FV, Heinrigs M, et al.: Phase III study evaluating the role of docetaxel in the adjuvant setting of breast cancer patients with = 4 involved lymph nodes: ADEBAR study. [Abstract] J Clin Oncol 23 (Suppl 16): A-908, 104s, 2005.
- [Result] Sommer HL, Janni W, Rack B, et al.: The ADEBAR-trial: the sequencing of regional radiotherapy and chemotherapy does not influence cytostatic dose intensity. [Abstract] J Clin Oncol 23 (Suppl 16): A-744, 64s, 2005.